CLINICAL TRIAL: NCT04189419
Title: A Phase 1/2a Clinical Trial to Evaluate the Efficacy and Safety of SCM-AGH in Patients With Moderate to Severe Acute Pancreatitis
Brief Title: Safety and Efficacy of SCM-AGH in Patients With Moderate to Severe Acute Pancreatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SCM Lifescience Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APT2001
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2022-05

CONDITIONS: Pancreatitis, Acute
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Intervention Model Description: Phase I: Multicenter in Korea, Non-Randomized, Open-label, Single arm, 3+3 design Phase II: Multicenter in Korea, Randomized, Double-blind, Placebo-controlled, 2-arm, Parallel Group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCM-AGH (Experimental): * Ingredient: Allogeneic human bone marrow derived mesenchymal stem cells
  * Dose: 1x10^6 cells/Kg
  Interventions: Biological: SCM-AGH
- Placebo (Placebo Comparator): IV infusion.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: SCM-AGH — SCM-AGH will be administrated once a day for 3 days(D0, D1 and D2).
  Arms: SCM-AGH
Other: Placebo — Placebo will be administrated once a day for 3 days(D0, D1 and D2).
  Arms: Placebo

SUMMARY:
This study consists of two phases (Phase I and Phase IIa). Phase IIa will be conducted sequentially after the safety of SCM-AGH is secured in Phase I.

* Phase I: Multicenter in Korea, Non-Randomized, Open-label, Single Arm, 3+3 design) for Severe Acute Pancreatitis
* Phase II: Multicenter in Korea, Randomized, Double-blind, 2-arm, Placebo-controlled, Parallel arm for Moderate to Severe Acute Pancreatitis

DETAILED DESCRIPTION:
Phase I (Multicenter in Korea, Non-Randomized, Open-label, Single Arm, 3+3 design): Three and up to six patients with severe Acute Pancreatitis are planned to recruit from 12 sites in Korea, but additional three patients can be enrolled by an assessment of Adverse Drug Reaction(ADR) from first three subjects .

Subjects will be administered with SCM-AGH as an intravenous (IV) infusion once a day for 3 days. Efficacy and safety are assessed daily for the first week, and then weekly on 3 occasions (Day 14, 21, and 28). Survival is followed up until Day 90.

Phase II (Multicenter in Korea, Randomized, Double-blind, 2-arm, Placebo-controlled, Parallel arm): Eligible patients will be randomized to the SCM-AGH group or placebo group at 1:1 ratio. Total 36 patients with Moderate to Severe Acute Pancreatitis are planned to be enrolled from 12 sites in Korea. Subjects will receive SCM-AGH on Day 0, 1, and 2. Existing standard of care is permitted. Efficacy and safety are assessed daily for the first week, and then weekly on 3 occasions (Day 14, 21, and 28). Survival is followed up until Day 90.

ELIGIBILITY:
Inclusion Criteria:

1. >=19 years of age

   [Phase I]
2. Patient with acute pancreatitis with organ failure which has been determined as severe acute pancreatitis prior to assignment(randomization) (1) Organ failure: 2 points of Modified Marshall Score in one or more of the respiratory system, renal system and cardiovascular system (2) Acute pancreatitis: at least 2 of the following 3 conditions are met

   1. Typical abdominal pain indicating acute pancreatitis
   2. Increased blood level of pancreatic enzyme (amylase or lipase >= three times of upper limit of normal)
   3. Finding acute pancreatitis in imaging test (contrast enhanced computerized tomography, abdominal magnetic resonance imaging, or abdominal sonography) (3) Severe: at least 1 of following organ failures lasting for > 48 hours according to the 2012 Atlanta Classification

      - Respiratory system: PaO2/FiO2 =< 300

      - Renal system: Creatinine >= 1.9 mg/dL
      * Cardiovascular system: low systolic blood pressure persists despite fluid replacement (SBP < 90 mmHg. off inotropic support)
3. Patient who or whose representative voluntarily agrees to participate in this study and has given a written informed consent

[Phase II] 2) Patient with acute pancreatitis with organ failure or CTSI score >= 4 which has been determined as moderate to severe acute pancreatitis prior to assignment(randomization)

1. Organ failure: 2 points of Modified Marshall Score in one or more of the respiratory system, renal system and cardiovascular system
2. CTSI: Sum of Balthazar grade and Necrosis score. CTSI 1-3: Mild / CTSI 4-6: Moderate / CTSI 7-10: Severe
3. Acute pancreatitis: at least 2 of the following 3 conditions are met

   a.Typical abdominal pain indicating acute pancreatitis b. Increased blood level of pancreatic enzyme (amylase or lipase >= three times of upper limit of normal) c. Finding acute pancreatitis in imaging test (contrast enhanced computerized tomography, abdominal magnetic resonance imaging, or abdominal sonography)
4. Moderate to Severe at least 1 of following organ failures lasting according to the 2012 Atlanta Classification - Respiratory system: PaO2/FiO2 =< 300 - Renal system: Creatinine >= 1.9 mg/dL

   * Cardiovascular system: low systolic blood pressure persists despite fluid replacement (SBP < 90 mmHg. off inotropic support)

[Moderately Severe]

* organ failures lasting for < 48 hours according to the 2012 Atlanta Classification or CTSI 4-8,

[Severe]

* organ failures lasting for >= 48 hours according to the 2012 Atlanta Classification

  3) Patient who or whose representative voluntarily agrees to participate in this study and has given a written informed consent

Exclusion Criteria:

1. Patient with allergic or hypersensitivity reaction to investigational product, drug of similar class or ingredients (bovine serum, dimethyl sulfoxide)
2. Patient who cannot undergo contrast-enhanced computerized tomography due to allergic reaction to contrast medium
3. Patient past >72 hours after the onset of organ failure at assignment (randomization)
4. Patient with condition that may develop acute abdominal pain
5. Patient with pancreatitis resulting from trauma, surgery, or neoplasm
6. Patient with unstable ventilation due to underlying disease other than pancreatitis
7. Patient with active infection such as non-pancreatic infection, septicemia, or pneumonia resulting from other disease
8. Patient requiring urgent surgery within 7 days
9. Patient with severe comorbidity (chronic renal disease, hepatic cirrhosis, chronic obstructive lung disease, bronchial asthma, congestive heart failure)
10. Patient with evidence of chronic pancreatitis (recurrent, obstructive and chronic; autoimmune and chronic; marked pancreatic insufficiency such as steatorrhea)
11. Pregnant woman, breastfeeding woman, or woman and man of reproductive potential not willing to use contraceptive measures during the study period
12. Patient who received other investigational product/device within 30 days prior to screening
13. Patient not eligible for study participation in the opinion of the investigator
14. Patient with current or past malignancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
The change from baseline in modified Marshall score on Day 7 for organ failure subject | Day 7
  The modified Marshall score is the scoring system to define the organ failure. The score is based on three different scores, one each for the respiratory, cardiovascular and renal. the modified Marshall score is >2 through the respiratory, renal or cardiovascular system, it is called organ failure.
The change from baseline in CTSI Score on Day 28 | Day 28 for CTSI Subject
  CTSI is scoring system to define the severity of acute pancreatitis. (4-6: Moderate, 7-10: Severe)

SECONDARY OUTCOMES:
Percentage of subjects whose organ failure was resolved at 3 days, 7 days, 14 days and 28 days | Day 3, Day 7, Day 14 and Day 28 or the day of discharge
The change from baseline in modified Marshall score at each assessment point up to Day 28 | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 14, Day 21, Day 28
The change from baseline in sequential organ failure assessment (SOFA) at each assessment point up to Day 28 | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 14, Day 21, Day 28 or the day of discharge
  SOFA score is used to track a person's status during the stay in an intensive care unit (ICU) to determine the extent of a person's organ function or rate of failure. The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems.
Duration of Systemic inflammatory response syndrome (SIRS) | Day 0, Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 14, Day 21, Day 28 or the day of discharge
Time to resolution of organ failure | Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 14, Day 21, Day 28
  The modified marshall score is 0 or 1 for all organ in respiratory, cardiovascular and renal.
The change from baseline value of C-Reactive Protein(CRP) which is inflammatory marker on Day 1, 2, 3, 5, 7, and 14 | Day 1, Day 2, Day 3, Day 5, Day 7, Day 14
Change from baseline in inflammatory markers(change of Tumor Necrosis Factor(TNF)-α, interleukin(IL)-6, TGF-b1, CCL2 and Lymphocyte count ratio) on Day 1, 2, 3, 5, 7, and 14 | Day 1, Day 2, Day 3, Day 5, Day 7, Day 14
Duration of intensive care unit (ICU) stay | Day 28 or the day of discharge
  Number of days for stay duration at ICU. The duration is from the day of hospitalization to day of discharge.
The change from baseline in Computed Tomography Severity Index(CTSI) on Day 28 | Day 28 or the day of discharge
  CTSI is the sum of Balthazar grade and necrosis score. The scoring is defined by evaluation of abdominal Computed Tomography(CT).
Incidence of pancreatic complication | Day 28 or the day of discharge
  Pancreatic complication will be evaluated by abdominal CT.
Requirement of drainage or surgery | Day 28 or the day of discharge
  Requirement of drainage due to intra-abdominal catastrophe or necrosis and surgery due to hemorrhage, perforation or abdominal compartment syndrome will be evaluated until Day 28.
Rate of infection | Day 28 or the day of discharge
  The even of infection such as infected pancreatic necrosis, bacteremia and pneumonia. The several tests for diagnosis can be conducted per investigator's decision.
Mortality on Day 28 and 90 | Day 28 or the day of discharge and Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Yun Nah Lee, Principal Investigator — Soon Chun Hyang University
Locations (7):
- South Korea (7):
  - Soonchunhyang University Hosptial Bucheon, Bucheon-si, Gyenggi-do
  - Kyungpook National University Chilgok Hospital, Daegu
  - Dongguk University Ilsan Hospital, Goyang-si
  - Chonnam National University Medical School, Gwangju
  - Inha University Hospital, Incheon
  - Ajou University Hospital, Suwon
  - Wonju Severance Christian Hospital, Wŏnju